CLINICAL TRIAL: NCT06420271
Title: Effects of Combined Transcranial Electrical and Magnetic Stimulation of Cerebellum on Balance Function in Ataxia Patients
Brief Title: Effects of Cerebellar tACS-iTBS in Ataxia
Acronym: EtABeta
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 80/SL/23
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-09

CONDITIONS: Ataxia
Keywords: Non Invasive Brain Stimulation; Transcranial Magnetic Stimulation; Intermittent Theta Burst Stimulation; Transcranial Electrical Stimulation; Transcranial Alternating Current Stimulation; Exergaming
MeSH Terms: conditions — Ataxia

STUDY DESIGN:
Intervention Model Description: A randomized cross-over design will be used. A 3-weeks wash-out period will be observed between the two conditions (real and sham).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tACS + real iTBS + exergaming (Experimental): 10 sessions of real 5Hz tACS with real iTBS + exergaming biofeedback, 5 times per weeks for two weeks.
  Interventions: Device: Real (real iTBS/tACS + exergaming)
- Sham tACS + sham iTBS + exergaming (Placebo Comparator): 10 sessions of sham 5Hz tACS with sham iTBS + exergaming biofeedback, 5 times per weeks for two weeks.
  Interventions: Device: Sham (sham iTBS/tACS + exergaming)

INTERVENTIONS:
Device: Real (real iTBS/tACS + exergaming) — Stimulation will be applied to the cerebellum. The tACS session duration will be 190 seconds with a frequency of 5 Hz coupled with iTBS (coil positioned tangentially with respect to the scalp)(600 pulses consisting of bursts of 3 stimuli at 50 Hz, repeated at intervals of 200ms, with an intensity of 80% of active motor threshold -AMT-) (Huang et al., 2005) for a total duration of 190 seconds. The exergaming will be performed with an adaptive system, comprising a force platform connected to a computer. The system is designed to enhance standard balance rehabilitation programs by guiding the user's performance of prescribed physical exercises through a video interface. Patients will perform 3 different exercises (10 minutes of training for a total of 30 minutes): 1) latero-lateral load shift; 2) antero posterior load shift; 3) omnidirectional displacement (combined latero-lateral and antero-posterior loading).
  Other Names: real iTBS/tACS + exergaming
  Arms: Real tACS + real iTBS + exergaming
Device: Sham (sham iTBS/tACS + exergaming) — Stimulation will be applied to the cerebellum. The tACS session duration will be 10 seconds with a frequency of 5 Hz coupled with sham iTBS (coil positioned perpendicularly with respect to the scalp)(600 pulses consisting of bursts of 3 stimuli at 50 Hz, repeated at intervals of 200ms, with an intensity of 80% of active motor threshold -AMT-) (Huang et al., 2005) for a total duration of 190 seconds. The exergaming will be performed with an adaptive system, comprising a force platform connected to a computer. The system is designed to enhance standard balance rehabilitation programs by guiding the user's performance of prescribed physical exercises through a video interface. Patients will perform 3 different exercises (10 minutes of training for a total of 30 minutes): 1) latero-lateral load shift; 2) antero posterior load shift; 3) omnidirectional displacement (combined latero-lateral and antero-posterior loading).
  Other Names: sham iTBS/tACS + exergaming
  Arms: Sham tACS + sham iTBS + exergaming

SUMMARY:
Ataxia refers to a group of neurological disorders characterized by impaired coordination and balance due to dysfunction in the cerebellum or its connections. Traditional therapeutic approaches for ataxia have shown limited efficacy, prompting researchers to explore alternative interventions. Non-invasive brain stimulation (NIBS) techniques, such as transcranial magnetic stimulation (TMS), transcranial direct current stimulation (tDCS), transcranial alternating current stimulation (tACS), and intermittent theta burst stimulation (iTBS), have emerged as potential therapeutic options. The aim of this study is to investigate the combined effect of tACS-iTBS on balance functions in ataxia disorders.

DETAILED DESCRIPTION:
Ataxia comprises a heterogeneous group of acquired or inherited disorders primarily involving cerebellar dysfunction, leading to impaired coordination and motor learning. Traditional treatments, including medication and physical therapy, often provide limited symptomatic improvement. Non-invasive brain stimulation (NIBS) techniques have emerged as promising tools for modulating cerebellar activity and enhancing motor function. Transcranial magnetic stimulation (TMS) can influence cortical excitability and plasticity, and studies have shown that high-frequency cerebellar rTMS can improve motor performance in spinocerebellar ataxia. Intermittent theta burst stimulation (iTBS), a patterned form of TMS, has demonstrated benefits in other movement disorders, suggesting potential applicability to ataxia. Transcranial direct current stimulation (tDCS), which modulates neuronal excitability via weak electrical currents, has shown improvements in static and dynamic balance in degenerative cerebellar ataxia. Transcranial alternating current stimulation (tACS) modulates neural oscillations and early studies indicate possible benefits for ataxia symptoms. Recent work has explored combining NIBS modalities to enhance neuromodulatory effects. In preliminary experiments, combined cerebellar tACS and iTBS increased MEP amplitudes more than iTBS alone, with effects lasting up to 30 minutes. These synergistic effects may translate into improved motor performance, coordination, and balance. The present study aims to investigate whether combining real or sham tACS with iTBS produces greater benefits than exergaming biofeedback alone in individuals with ataxia. A cross-over design will be used so that each participant serves as their own control. The primary outcomes will include motor coordination, balance, and cerebello-cortical plasticity. The rationale is that tACS may optimize oscillatory activity while iTBS enhances excitability, thereby jointly promoting neuroplasticity in cerebellar networks. The study will recruit individuals diagnosed with ataxia and assess the therapeutic potential of combined NIBS interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of ataxia based on clinical assessment and/or neuroimaging findings.
2. Stable medication regimen for at least four weeks prior to the study.
3. Sufficient cognitive ability to understand and comply with study instructions.

Exclusion Criteria:

1. History of seizures.
2. Severe general impairment or concomitant diseases.
3. Intracranial metal implants.
4. Cardiac pacemaker.
5. Pregnancy status.

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the International Cooperative Ataxia Rating Scale (ICARS) | Baseline (1), 2 weeks from baseline (1), Baseline (2), 2 weeks from baseline (2)
  ICARS was developed to quantify the level of impairment as a result of ataxia as related to hereditary ataxias. Score ranges from 0 to 100 where 100 indicates severe ataxia.

SECONDARY OUTCOMES:
Changes in the Short Form-36 Health Survey (SF-36) | Baseline (1), 2 weeks from baseline (1), Baseline (2), 2 weeks from baseline (2)
  SF-36 is an outcome measure instrument that is often used, well-researched, self-reported measure of health. Scores range from 0 to 100 for each domain, where 100 indicates a more favorable health-state.
Changes in postural control | Baseline (1), 2 weeks from baseline (1), Baseline (2), 2 weeks from baseline (2)
  Instrumented postural stability will be assessed using a 75 cm (length x width) static force platform (PlatformBPM 120, Physical Support Italia, Italy). The signals will be amplified and acquired using dedicated software (Physical Gait Software Vv. 2.66, Physical SupportItalia, Italy). The length of the center of pressure (CoP) trajectory (mm) will be measured as indicator of the postural stability. An increase in the length of CoP indicates a severe impairment in postural control.
Changes in cortico-spinal excitability | Baseline (1), 2 weeks from baseline (1), Baseline (2), 2 weeks from baseline (2)
  Twenty Motor evoked potentials (MEPs) will be collected from left and right primary motor cortex with single pulses of transcranial magnetic stimulation (TMS) set at 1 mV. An increase in the MEPs amplitude indicates an improvement in cortico-spinal activity recorded from the first dorsal interosseous and tibialis anterior muscles.
Change in the Scale for the Assessment and Rating of Ataxia (SARA) | Baseline (1), 2 weeks from baseline (1), Baseline (2), 2 weeks from baseline (2)
  SARA is a clinical scale developed to assess a range of different impairments in cerebellar ataxia. The scale is made up of 8 items related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements and heel-shin test. Score ranges from 0 to 40 where 40 indicates severe ataxia.

OTHER OUTCOMES:
Change in Cerebellar Brain Inhibition (CBI) | Baseline (1), 2 weeks from baseline (1), Baseline (2), 2 weeks from baseline (2)
  CBI will be performed with two Magstim figure-of-eight coils (70 mm diameter), one placed over the primary motor cortex and the other centered over the contralateral cerebellar hemisphere, 3 cm lateral to the Inion with an upward current induced to the brain. For each CBI evaluation, we will record 20 TMS test stimuli (TS) over the M1 that were set at intensity to elicit an MEP ∼1 mV. In half of these trials, selected randomly, a TMS conditioning stimulus (CS) was delivered over the contralateral cerebellar hemisphere 5 ms prior to the TS at an intensity of 120% of the resting motor threshold (RMT). Thus, a total of 20 TS and 20 CS + TS pulses will be administered. CBI will be calculated as the ratio of the mean MEP amplitude in the CS + TS relative to TS. An increase in CBI indicates higher connectivity between the cerebellum and primary motor cortex.

CONTACTS AND LOCATIONS:
Overall Officials: Danny Spampinato, PhD, Study Chair — University of Roma La Sapienza; Alex Martino Cinnera, PhD, Study Chair — IRCCS Santa Lucia Foundation
Locations (1):
- IRCCS Santa Lucia Foundation, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spampinato D, Avci E, Rothwell J, Rocchi L. Frequency-dependent modulation of cerebellar excitability during the application of non-invasive alternating current stimulation. Brain Stimul. 2021 Mar-Apr;14(2):277-283. doi: 10.1016/j.brs.2021.01.007. Epub 2021 Jan 20. PMID 33482375
- [Background] Libri I, Cantoni V, Benussi A, Rivolta J, Ferrari C, Fancellu R, Synofzik M, Alberici A, Padovani A, Borroni B. Comparing Cerebellar tDCS and Cerebellar tACS in Neurodegenerative Ataxias Using Wearable Sensors: A Randomized, Double-Blind, Sham-Controlled, Triple-Crossover Trial. Cerebellum. 2024 Apr;23(2):570-578. doi: 10.1007/s12311-023-01578-6. Epub 2023 Jun 22. PMID 37349632
- [Background] Guerra A, Suppa A, Bologna M, D'Onofrio V, Bianchini E, Brown P, Di Lazzaro V, Berardelli A. Boosting the LTP-like plasticity effect of intermittent theta-burst stimulation using gamma transcranial alternating current stimulation. Brain Stimul. 2018 Jul-Aug;11(4):734-742. doi: 10.1016/j.brs.2018.03.015. Epub 2018 Mar 24. PMID 29615367
- [Background] Gong C, Long Y, Peng XM, Hu H, Chen J, Xiao L, Zhong YB, Wang MY, Luo Y. Efficacy and safety of noninvasive brain stimulation for patients with cerebellar ataxia: a systematic review and meta-analysis of randomized controlled trials. J Neurol. 2023 Oct;270(10):4782-4799. doi: 10.1007/s00415-023-11799-8. Epub 2023 Jul 17. PMID 37460852